CLINICAL TRIAL: NCT00716274
Title: Neurophysiology of Attention-Deficit/Hyperactivity Disorder (ADHD) and Comorbid Dyslexia: Functional Magnetic Resonance Imaging (fMRI) Measures of Brain Activation During Attention and Reading Tasks Pre- and Post-Atomoxetine Treatment
Brief Title: Effects of Atomoxetine on Brain Activation During Attention & Reading Tasks in Participants With ADHD & Comorbid Dyslexia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12212; B4Z-US-LYEI (Other: Eli Lilly and Company); 2019-000419-98 (EudraCT Number)
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Attention Deficit Hyperactivity Disorder; Dyslexia
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Dyslexia | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Experimental): Atomoxetine will be administered at 1.0 to 1.4 mg/kg/day given orally once daily in the morning for 16 weeks (study period II). Participants who complete the study period II will be re-randomized in the study period III of 16-week duration to assess maintenance of benefit following discontinuation of treatment with atomoxetine. Participants assigned to atomoxetine during the study period II will be re-randomized to either atomoxetine or placebo whereas participants previously assigned to placebo will receive atomoxetine.
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Placebo will be packaged in the same way as active comparator to enforce double-blind study design
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Atomoxetine will be administered at 1.0 to 1.4 mg/kg/day given orally once daily in the morning for 16 weeks
  Other Names: LY139603
  Arms: Atomoxetine
Drug: Placebo — oral, daily, for 16 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate the effects of atomoxetine on brain activation during attention and reading tasks via functional Magnetic Resonance Imaging (fMRI) in participants ages 10 to 16 years old with ADHD and comorbid dyslexia

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, single site study that uses an fMRI measurement to assess brain activation during attention and reading tasks and the effects of atomoxetine in reducing symptoms of ADHD in participants with ADHD and comorbid dyslexia. Similar assessments are performed in two additional groups of participants with ADHD only and dyslexia only to determine to what extent symptomatic change in the comorbid ADHD & dyslexia is achieved independently by atomoxetine effects on either condition. A healthy control group of non-ADHD, non-dyslexia subjects (20) will be included to monitor practice effects & effects of treatment that may be interpreted as normal maturation. The healthy control group will not be treated with any study medications.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the ADHD-only or ADHD+dyslexia groups must meet DSM-IV-TR criteria for ADHD
* Participants in the dyslexia-alone group or ADHD+dyslexia groups must meet criteria for dyslexia
* Participants must achieve a score of 80 or more on the Full Scale Intelligence Quotient
* Child or adolescent participants must be 10 to 16 years old
* Must be able to communicate in English
* Must be able to swallow capsules
* Be reliable to keep appointments for clinic visits & all related tests
* Participants for healthy control group do not meet DSM-IV-TR criteria for ADHD and/or dyslexia
* Participants for healthy control group must achieve a score of at least 80 but not >120 on the Full Scale Intelligence Quotient

Exclusion Criteria:

* Participants who weigh less than 25.1 kilogram (kg) or greater than 70 kg.
* Participants with severe allergies to more than 1 class of medications or who have had multiple adverse drug reactions
* Participants with prior diagnosis of bipolar I or bipolar II disorder or psychosis
* Participants with documented history of autism, Asperger's syndrome, or pervasive developmental disorder
* Females who are pregnant or breastfeeding
* Participants treated with atomoxetine at a therapeutic dose (1.2 mg/kg/day) for at least 4 to 6 weeks

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2008-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to either atomoxetine or placebo during study period II. Placebo participants were then assigned to atomoxetine in study period III. Atomoxetine participants were re-randomized to atomoxetine or placebo in study period III. Participants assigned to the healthy control group did not receive any study drug.
Groups:
- Atomoxetine: Atomoxetine (ATX) 1.0 to 1.4 milligram/kilogram/day (mg/kg/day) was administered orally once daily in the morning for 16 weeks, during study period II, (SP II). All eligible participants who received atomoxetine during study period II and completed that period were re-randomized to atomoxetine or placebo in study period III (SP III).
- Placebo: Placebo (PLA) was packaged in the same way as active comparator to enforce double-blind study design. Placebo was given orally, daily for 16 weeks during SP II. All eligible participants who received placebo during SP II and completed that period were assigned atomoxetine in SP III.
- ATX/ATX: These participants were randomized to atomoxetine in SP II and were re-randomized to atomoxetine in SP III. Atomoxetine was dosed orally once-daily in the morning 0.5 mg/kg/day for 3 days and then titrated up to a dose between 1.2 and 1.4 mg/kg/day.
- ATX/PLA: These participants were randomized to atomoxetine in SP II and were re-randomized to placebo in SP III. Atomoxetine was dosed orally once-daily in the morning 0.5 mg/kg/day for 3 days and then titrated up to a dose between 1.2 and 1.4 mg/kg/day.
- PLA/ATX: These participants were randomized to placebo in SP II and were assigned to atomoxetine in SP III. Atomoxetine was dosed orally once-daily in the morning 0.5 mg/kg/day for 3 days and then titrated up to a dose between 1.2 and 1.4 mg/kg/day.
- Healthy Participants: Healthy Participants: Participants were evaluated to confirm that they did not meet criteria for Attention Deficit Hyperactivity Disorder (ADHD) or dyslexia. They received no treatment during the study.
Period: Study Period II (16-Weeks)
Arm/Group | Atomoxetine | Placebo | ATX/ATX | ATX/PLA | PLA/ATX | Healthy Participants
Started | 45 | 44 | 0 | 0 | 0 | 21
Completed | 36 | 35 | 0 | 0 | 0 | 19
Not Completed | 9 | 9 | 0 | 0 | 0 | 2
Not completed — Entry Criteria Not Met | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 3 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 1 | 0 | 0 | 0 | 1
Not completed — Parent/Caregiver Decision | 3 | 3 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0 | 0
Period: Study Period III (16-Weeks)
Arm/Group | Atomoxetine | Placebo | ATX/ATX | ATX/PLA | PLA/ATX | Healthy Participants
Started | 0 (Participants were assessed for maintenance of benefit after discontinuation of atomoxetine.) | 0 (Participants were assessed for maintenance of benefit after discontinuation of atomoxetine.) | 18 (Participants were assessed for maintenance of benefit after discontinuation of atomoxetine.) | 18 (Participants were assessed for maintenance of benefit after discontinuation of atomoxetine.) | 35 (Participants were assessed for maintenance of benefit after discontinuation of atomoxetine.) | 19 (Participants were assessed for maintenance of benefit after discontinuation of atomoxetine.)
Completed | 0 | 0 | 16 | 17 | 32 | 19
Not Completed | 0 | 0 | 2 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Parent Caregiver Decision | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atomoxetine: Atomoxetine 1.0 to 1.4 mg/kg/day was administered orally once daily in the morning for 16 weeks, during SP II. All eligible participants who received atomoxetine during SP II and completed that period were re-randomized to atomoxetine or placebo in SP III.
- Placebo: Placebo was packaged in the same way as active comparator to enforce double-blind study design. Placebo was given orally, daily for 16 weeks during SP II. All eligible participants who received placebo during SP II and completed that period were assigned atomoxetine in SP III.
- Healthy Participants: Healthy Participants: Participants were evaluated to confirm that they did not meet criteria for ADHD or dyslexia. They received no treatment during the study.
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Healthy Participants | Total
Number analyzed (Participants) | 45 | 44 | 21 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (1.89) | 12.1 (1.90) | 12.4 (2.05) | 12.20 (1.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 13 | 48
  Male | 27 | 27 | 8 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 4 | 12
  Not Hispanic or Latino | 39 | 42 | 17 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 13 | 5 | 22
  White | 33 | 29 | 12 | 74
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 2 | 4 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 44 | 21 | 110

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint in Functional Magnetic Resonance Imaging (fMRI) Activation in Participants With Dyslexia Alone (Pseudoword Rhyming and Semantic-category)
Description: Change From Baseline in Task-related Brain Activity During Biological Motion Recognition Task (Task-based fMRI) BOLD response (Blood-oxygen-level-dependent response)
Time Frame: Baseline, 16 Weeks
Population: All participants who received study drug, had Dyslexia Alone and had fMRI data.
Measure: Mean (Standard Deviation); unit: Change-from-baseline (BOLD response)
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 13 | 10
Change-from-baseline (BOLD response)
  Semantic-category: Left Inferior Frontal Gyrus | -0.056 (0.125) | -0.033 (0.118)
  Semantic-category: Left Interior Temporal Gyrus | -0.061 (0.120) | 0.010 (0.075)
  Semantic-category: Left Medial Temporal Gyrus | -0.038 (0.153) | -0.006 (0.053)
  Semantic-category: Left Temporo-parietal Region | -0.073 (0.124) | -0.037 (0.100)
  Semantic-category: Right Inferior Frontal Gyrus | 0.019 (0.156) | 0.018 (0.147)
  Semantic-category: Right Interior Temporal Gyrus | 0.002 (0.217) | 0.058 (0.161)
  Semantic-category: Right Medial Temporal Gyrus | -0.014 (0.181) | 0.071 (0.091)
  Semantic-category: Right Temporo-parietal Region | -0.015 (0.145) | 0.076 (0.114)
  Pseudoword Rhyming: Left Inferior Frontal Gyrus: number analyzed (Participants) | 13 | 9
  Pseudoword Rhyming: Left Inferior Frontal Gyrus | 0.012 (0.200) | 0.020 (0.147)
  Pseudoword Rhyming: Left Interior Temporal Gyrus: number analyzed (Participants) | 13 | 9
  Pseudoword Rhyming: Left Interior Temporal Gyrus | -0.062 (0.200) | -0.003 (0.109)
  Pseudoword Rhyming: Left Medial Temporal Gyrus: number analyzed (Participants) | 13 | 9
  Pseudoword Rhyming: Left Medial Temporal Gyrus | 0.005 (0.253) | 0.024 (0.133)
  Pseudoword Rhyming: Left Temporo-parietal Region: number analyzed (Participants) | 13 | 9
  Pseudoword Rhyming: Left Temporo-parietal Region | -0.026 (0.243) | -0.012 (0.115)
  Pseudoword Rhyming: Right Inferior Frontal Gyrus: number analyzed (Participants) | 13 | 9
  Pseudoword Rhyming: Right Inferior Frontal Gyrus | -0.017 (0.304) | 0.024 (0.187)
  Pseudoword Rhyming: Right Interior Temporal Gyrus: number analyzed (Participants) | 13 | 9
  Pseudoword Rhyming: Right Interior Temporal Gyrus | 0.013 (0.266) | 0.103 (0.174)
  Pseudoword Rhyming: Right Medial Temporal Gyrus: number analyzed (Participants) | 13 | 9
  Pseudoword Rhyming: Right Medial Temporal Gyrus | 0.039 (0.250) | 0.009 (0.098)
  Pseudoword Rhyming: Temporo-parietal Region: number analyzed (Participants) | 13 | 9
  Pseudoword Rhyming: Temporo-parietal Region | 0.011 (0.296) | 0.087 (0.170)

2. Primary Outcome: Change From Baseline to Endpoint in fMRI Activation in Participants With Dyslexia Alone (Stroop Attention Tasks)
Description: Change From Baseline to Endpoint in fMRI Activation in Participants With Dyslexia Alone (Stroop Attention Tasks)
Time Frame: Baseline, 16 Weeks
Population: Stroop Tasks data were not collected.
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change From Baseline to Endpoint in fMRI Activation in Participants With ADHD or ADHD + Dyslexia (Pseudoword Rhyming and Semantic-category Tasks)
Description: as for outcome 1
Time Frame: Baseline, 16 Weeks
Population: All participants who received study drug, had ADHD or ADHD + Dyslexia and had fMRI data.
Measure: Mean (Standard Deviation); unit: Change-from-baseline (BOLD response)
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 11 | 12
Change-from-baseline (BOLD response)
  ADHD+Dyslexia, Semantic-category: Left Inferior Frontal Gyrus: number analyzed (Participants) | 10 | 12
  ADHD+Dyslexia, Semantic-category: Left Inferior Frontal Gyrus | 0.077 (0.085) | -0.038 (0.141)
  ADHD+Dyslexia, Semantic-category: Left Interior Temporal Gyrus: number analyzed (Participants) | 10 | 12
  ADHD+Dyslexia, Semantic-category: Left Interior Temporal Gyrus | 0.079 (0.128) | -0.1 (0.252)
  ADHD+Dyslexia, Semantic-category: Left Medial Temporal Gyrus: number analyzed (Participants) | 10 | 12
  ADHD+Dyslexia, Semantic-category: Left Medial Temporal Gyrus | 0.038 (0.105) | -0.037 (0.208)
  ADHD+Dyslexia, Semantic-category: Left Temporo-parietal Region: number analyzed (Participants) | 10 | 12
  ADHD+Dyslexia, Semantic-category: Left Temporo-parietal Region | 0.079 (0.065) | -0.096 (0.187)
  ADHD+Dyslexia, Semantic-category: Right Inferior Frontal Gyrus: number analyzed (Participants) | 10 | 12
  ADHD+Dyslexia, Semantic-category: Right Inferior Frontal Gyrus | 0.065 (0.095) | -0.016 (0.152)
  ADHD+Dyslexia, Semantic-category: Right Interior Temporal Gyrus: number analyzed (Participants) | 10 | 12
  ADHD+Dyslexia, Semantic-category: Right Interior Temporal Gyrus | 0.008 (0.150) | 0.015 (0.222)
  ADHD+Dyslexia, Semantic-category: Right Medial Temporal Gyrus: number analyzed (Participants) | 10 | 12
  ADHD+Dyslexia, Semantic-category: Right Medial Temporal Gyrus | -0.046 (0.169) | -0.045 (0.168)
  ADHD+Dyslexia, Semantic-category: Right Temporo-parietal Region: number analyzed (Participants) | 10 | 12
  ADHD+Dyslexia, Semantic-category: Right Temporo-parietal Region | 0.053 (0.120) | -0.035 (0.153)
  ADHD+Dyslexia, Pseudoword Rhyming: Left Inferior Frontal Gyrus: number analyzed (Participants) | 9 | 11
  ADHD+Dyslexia, Pseudoword Rhyming: Left Inferior Frontal Gyrus | 0.081 (0.245) | 0.005 (0.151)
  ADHD+Dyslexia, Pseudoword Rhyming: Left Interior Temporal Gyrus: number analyzed (Participants) | 9 | 11
  ADHD+Dyslexia, Pseudoword Rhyming: Left Interior Temporal Gyrus | 0.142 (0.370) | 0.047 (0.202)
  ADHD+Dyslexia, Pseudoword Rhyming: Left Medial Temporal Gyrus: number analyzed (Participants) | 9 | 11
  ADHD+Dyslexia, Pseudoword Rhyming: Left Medial Temporal Gyrus | 0.091 (0.387) | 0.042 (0.184)
  ADHD+Dyslexia, Pseudoword Rhyming: Left Temporo-parietal Region: number analyzed (Participants) | 9 | 11
  ADHD+Dyslexia, Pseudoword Rhyming: Left Temporo-parietal Region | 0.096 (0.321) | 0.012 (0.184)
  ADHD+Dyslexia, Pseudoword Rhyming: Right Inferior Frontal Gyrus: number analyzed (Participants) | 9 | 11
  ADHD+Dyslexia, Pseudoword Rhyming: Right Inferior Frontal Gyrus | 0.069 (0.291) | -0.006 (0.111)
  ADHD+Dyslexia, Pseudoword Rhyming: Right Interior Temporal Gyrus: number analyzed (Participants) | 9 | 11
  ADHD+Dyslexia, Pseudoword Rhyming: Right Interior Temporal Gyrus | 0.114 (0.453) | 0.047 (0.164)
  ADHD+Dyslexia, Pseudoword Rhyming: Right Medial Temporal Gyrus: number analyzed (Participants) | 9 | 11
  ADHD+Dyslexia, Pseudoword Rhyming: Right Medial Temporal Gyrus | 0.080 (0.470) | 0.002 (0.203)
  ADHD+Dyslexia, Pseudoword Rhyming: Temporo-parietal Region: number analyzed (Participants) | 9 | 11
  ADHD+Dyslexia, Pseudoword Rhyming: Temporo-parietal Region | 0.078 (0.308) | -0.026 (0.147)
  ADHD Only, Semantic-category: Left Inferior Frontal Gyrus: number analyzed (Participants) | 11 | 8
  ADHD Only, Semantic-category: Left Inferior Frontal Gyrus | 0.013 (0.166) | -0.057 (0.120)
  ADHD Only, Semantic-category: Left Interior Temporal Gyrus: number analyzed (Participants) | 11 | 8
  ADHD Only, Semantic-category: Left Interior Temporal Gyrus | -0.024 (0.083) | -0.035 (0.105)
  ADHD Only, Semantic-category: Left Medial Temporal Gyrus: number analyzed (Participants) | 11 | 8
  ADHD Only, Semantic-category: Left Medial Temporal Gyrus | -0.002 (0.168) | -0.047 (0.166)
  ADHD Only, Semantic-category: Left Temporo-parietal Region: number analyzed (Participants) | 11 | 8
  ADHD Only, Semantic-category: Left Temporo-parietal Region | -0.013 (0.131) | -0.064 (0.124)
  ADHD Only, Semantic-category: Right Inferior Frontal Gyrus: number analyzed (Participants) | 11 | 8
  ADHD Only, Semantic-category: Right Inferior Frontal Gyrus | -0.074 (0.141) | -0.030 (0.211)
  ADHD Only, Semantic-category: Right Interior Temporal Gyrus: number analyzed (Participants) | 11 | 8
  ADHD Only, Semantic-category: Right Interior Temporal Gyrus | 0.052 (0.236) | -0.100 (0.141)
  ADHD Only, Semantic-category: Right Medial Temporal Gyrus: number analyzed (Participants) | 11 | 8
  ADHD Only, Semantic-category: Right Medial Temporal Gyrus | -0.039 (0.240) | 0.019 (0.211)
  ADHD Only, Semantic-category: Right Temporo-parietal Region: number analyzed (Participants) | 11 | 8
  ADHD Only, Semantic-category: Right Temporo-parietal Region | 0.034 (0.124) | -0.101 (0.129)
  ADHD Only, Pseudoword Rhyming: Left Inferior Frontal Gyrus: number analyzed (Participants) | 11 | 8
  ADHD Only, Pseudoword Rhyming: Left Inferior Frontal Gyrus | -0.029 (0.153) | 0.101 (0.203)
  ADHD Only, Pseudoword Rhyming: Left Interior Temporal Gyrus: number analyzed (Participants) | 11 | 8
  ADHD Only, Pseudoword Rhyming: Left Interior Temporal Gyrus | -0.012 (0.194) | 0.063 (0.240)
  ADHD Only, Pseudoword Rhyming: Left Medial Temporal Gyrus: number analyzed (Participants) | 11 | 8
  ADHD Only, Pseudoword Rhyming: Left Medial Temporal Gyrus | -0.030 (0.137) | 0.058 (0.260)
  ADHD Only, Pseudoword Rhyming: Left Temporo-parietal Region: number analyzed (Participants) | 11 | 8
  ADHD Only, Pseudoword Rhyming: Left Temporo-parietal Region | -0.013 (0.172) | 0.029 (0.195)
  ADHD Only, Pseudoword Rhyming: Right Inferior Frontal Gyrus: number analyzed (Participants) | 11 | 8
  ADHD Only, Pseudoword Rhyming: Right Inferior Frontal Gyrus | 0.005 (0.139) | 0.088 (0.289)
  ADHD Only, Pseudoword Rhyming: Right Interior Temporal Gyrus: number analyzed (Participants) | 11 | 8
  ADHD Only, Pseudoword Rhyming: Right Interior Temporal Gyrus | -0.003 (0.226) | 0.043 (0.246)
  ADHD Only, Pseudoword Rhyming: Right Medial Temporal Gyrus: number analyzed (Participants) | 11 | 8
  ADHD Only, Pseudoword Rhyming: Right Medial Temporal Gyrus | 0.007 (0.116) | -0.011 (0.402)
  ADHD Only, Pseudoword Rhyming: Temporo-parietal Region: number analyzed (Participants) | 11 | 8
  ADHD Only, Pseudoword Rhyming: Temporo-parietal Region | -0.016 (0.204) | 0.046 (0.149)

4. Primary Outcome: Change From Baseline to Endpoint in fMRI Activation in Participants With ADHD or ADHD + Dyslexia (Stroop Tasks)
Description: Change From Baseline to Endpoint in fMRI Activation in Participants With ADHD or ADHD + Dyslexia (Stroop Tasks)
Time Frame: Baseline, 16 Weeks
Population: Stroop Tasks data were not collected.
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Change From Baseline to Endpoint in Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version (ADHDRS) Total Score in the ADHD or ADHD + Dyslexia
Description: The ADHDRS-IV-Parent is an 18-item scale with 1 item for each of the 18 symptoms contained in the DSM-IV diagnosis of ADHD. Each item is scored on a 0 to 3 scale: 0=none (never or rarely); 1=mild (sometimes); 2=moderate (often); 3=severe (very often). Total scores range from 0-54. Higher scores indicate higher impairment and lower scores indicate no impairment. LS mean was calculated using a restricted maximum likelihood (REML)-based, MMRM analysis which includes treatment, baseline, visit, treatment-by-visit interaction, and baseline-by-visit interaction.
Time Frame: Baseline, 16 weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post baseline ADHDRS-IV-Parent: Inv measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 23 | 23
units on a scale
  ADHD + Dyslexia: number analyzed (Participants) | 11 | 14
  ADHD + Dyslexia | -11.04 (2.518) | -7.53 (2.155)
  ADHD Alone: number analyzed (Participants) | 12 | 9
  ADHD Alone | -13.85 (2.323) | -1.63 (2.588)

6. Primary Outcome: Change From Baseline to Endpoint in Woodcock Johnson Tests of Achievement (WJ III) Word Attack Total Score in Participants With Dyslexia Alone
Description: WJ III (Woodcock et al. 2001) has two parallel forms (A and B) alternating two batteries of tests-Standard and Extended. Standard tests (1 -12) have a broad set of scores. Extended tests (13 -22) have a more in-depth diagnostic assessment of academic strengths and weaknesses. Tests administered were 1, 2, 7, 9, 13, 17, and 20. The standard score scale is a mean (M) of 100 and a standard deviation (SD) of 15. The WJ III ACH has extended standard scores which is a greater range of standard scores. Test 13, Word Attack, measures skill in applying phonic, structural analysis to the pronunciation of unfamiliar printed words. Each individual test scores range from 0 to over 200 where 69 and below is very low and 131 and above is very superior. Higher scores indicate better reading skills. Least Square (LS) Mean was analyzed using last observation carried forward (LOCF), fixed-effects analysis of covariate (ANCOVA) models with terms for treatment, gender, baseline, age, treatment*baseline.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post baseline WJ III measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale | -3.57 (4.84) | 2.92 (4.75)

7. Secondary Outcome: Change From Baseline to Endpoint in Basic Reading Skills Cluster WJ III in Participants With Dyslexia Alone
Description: WJ III (Woodcock et al. 2001) has two parallel forms (A and B) alternating two batteries of tests-Standard and Extended. The standard score scale is a mean (M) of 100 and a standard deviation (SD) of 15. Basic Reading Skills is an aggregate measure of sight vocabulary, phonics, and structural analysis. It is a combination of Test 1, Letter-Word Identification, which measures the participant's word identification skills, and Test 13, Word Attack, which measures skill in applying phonic and structural analysis skills to the pronunciation of unfamiliar printed words. It is the average (arithmetic mean) of the tests 1 and 13. Scores for each individual test range from 0 to over 200 where 69 and below is very low and 131 and above is very superior. Higher scores indicate better reading skills. LS mean was analyzed using LOCF, fixed-effects ANCOVA models with terms for treatment, gender, baseline, age, treatment*baseline.
Time Frame: Baseline, 16 Weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale | -2.81 (3.87) | 2.25 (3.85)

8. Secondary Outcome: Change From Baseline to Endpoint in BADD-A Total Score in Participants With ADHD or ADHD + Dyslexia
Description: The BADD-A is used to assess impairment in executive functions related to ADHD. These include 1) Organizing, prioritizing, and activating to work; 2) Focusing, sustaining and shifting attention to tasks; 3) Regulating alertness, sustaining effort, and processing speed; 4) Managing frustration and modulating emotions; 5) Utilizing working memory and accessing recall (Brown 2001). Scores range from 0-120. The higher the score the more severe the attention-deficit disorder (ADD). 0-39 equate to, "ADD possible but not likely". 40-54 equate to, "ADD probable but not certain". 55-120 equate to, "ADD highly probable". LS mean was calculated using a REML-based, MMRM analysis which includes treatment, baseline, visit, treatment-by-visit interaction, and baseline-by-visit interaction.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post baseline BADD-A measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 23 | 22
units on a scale
  ADHD + Dyslexia: number analyzed (Participants) | 11 | 14
  ADHD + Dyslexia | -6.91 (4.689) | -4.29 (4.128)
  ADHD Alone: number analyzed (Participants) | 12 | 8
  ADHD Alone | -9.05 (5.515) | -1.85 (6.695)

9. Secondary Outcome: Change From Baseline to Endpoint in WJ III Individual Test Scores in Participants With Dyslexia Alone
Description: WJ III (Woodcock et al. 2001) has two parallel forms (A and B) alternating two batteries of tests-Standard and Extended. Standard tests (1 -12) have a broad set of scores. Extended tests (13 -22) have a more in-depth diagnostic assessment of academic strengths and weaknesses. Tests administered were 1, 2, 7, 9, 13, 17, and 20. The standard score scale is a mean (M) of 100 and a standard deviation (SD) of 15. The WJ III ACH has extended standard scores, which is a greater range of standard scores. Scores for each individual test range from 0 to over 200 where 69 and below is very low and 131 and above is very superior. Higher scores indicate better reading skills. LS mean was analyzed using LOCF, fixed-effects ANCOVA models with terms for treatment, gender, baseline, age, treatment*baseline.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants who had a WJ III baseline and post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  Letter Word Identification | 0.88 (1.12) | 2.77 (1.10)
  Word Attack Score | 0.48 (1.71) | 2.53 (1.68)
  Reading Vocabulary Score | 1.04 (1.81) | -1.73 (1.75)
  Reading Fluency Score | 0.13 (1.59) | -1.06 (1.53)
  Reading Comprehension Score | 2.38 (1.81) | -1.03 (1.74)
  Spelling Score | 0.89 (1.50) | -0.36 (1.48)
  Spelling of Sounds Score | 3.11 (1.48) | 3.59 (1.43)
  Basic Reading Skills Score | 0.99 (1.15) | 2.13 (1.15)
  Passage Comprehension | 2.80 (2.03) | -0.20 (1.96)

10. Secondary Outcome: Change From Baseline to Endpoint in WJ III Individual Test Scores in Participants With ADHD + Dyslexia
Description: as for outcome 9
Time Frame: Baseline, 16 Weeks
Population: All randomized participants who had a baseline and post-baseline WJ III measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  Reading Fluency | -3.41 (2.16) | 2.61 (2.06)
  Reading Comprehension | 2.02 (1.63) | 0.80 (1.56)
  Letter Word Identification | 1.71 (1.75) | -0.90 (1.69)
  Word Attack Score | 2.65 (1.13) | 0.71 (1.07)
  Reading Vocabulary | 0.69 (1.89) | 2.80 (1.77)
  Spelling | -1.36 (2.25) | -2.59 (2.19)
  Spelling of Sounds | 8.42 (1.76) | 5.02 (1.67)
  Basic Reading Skills | 2.53 (1.05) | -0.21 (1.01)
  Passage Comprehension Score | 2.65 (1.71) | -1.01 (1.65)

11. Secondary Outcome: Change From Baseline to Endpoint in WJ III Individual Test Scores in Participants With ADHD Alone
Description: as for outcome 9
Time Frame: Baseline, 16 Weeks
Population: All randomized participants who had a baseline and post-baseline WJ III measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  Reading Fluency | -2.70 (1.58) | -4.98 (1.81)
  Reading Comprehension | -2.92 (2.39) | -1.40 (2.77)
  Letter Word Identification | 2.60 (1.77) | 0.46 (2.08)
  Word Attack Score | -1.60 (1.56) | 0.08 (1.78)
  Reading Vocabulary | -1.15 (2.65) | -1.48 (3.23)
  Spelling | 4.30 (1.20) | 3.62 (1.39)
  Spelling of Sounds | 5.90 (3.51) | 0.57 (4.04)
  Basic Reading Skills | 0.86 (1.42) | 0.48 (1.65)
  Passage Comprehension Score | -4.10 (2.36) | -1.80 (2.70)

12. Secondary Outcome: Change From Baseline to Endpoint in Comprehensive Test of Phonological Processing (CTOPP) Composite Scores in Participants With Dyslexia Alone
Description: The CTOPP assesses phonological awareness, phonological memory, and rapid naming and is appropriate for ages 7 to 24. The test contains six core subtests. The composite scores are 1) Phonological Awareness, comprised of the standard scores of the Elision and Blending Words; 2) Phonological Memory, comprised of standard scores for Memory for Digits and Non-word Repetition; and 3) Rapid Naming, comprised of standard scores for Rapid Digit Naming and Rapid Letter Naming. Standard scores range from 1-20, and composite scores range from 35-165. Higher scores are better and lower scores are poor. LS mean was analyzed using LOCF, fixed-effects ANCOVA models with terms for treatment, gender, baseline, age, treatment*baseline.
Time Frame: Baseline, 16 weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post baseline CTOPP measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 13 | 13
units on a scale
  Phonological Awareness | 4.01 (4.81) | 2.69 (1.91)
  Phonological Memory | 5.62 (1.82) | 0.62 (1.75)
  Rapid Naming Score | 0.19 (2.31) | -1.00 (2.23)

13. Secondary Outcome: Change From Baseline to Endpoint in CTOPP Composite Score in Participants With ADHD + Dyslexia
Description: as for outcome 12
Time Frame: Baseline, 16 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 12 | 15
units on a scale
  Phonological Awareness | 4.60 (1.74) | 1.35 (1.66)
  Phonological Memory | 2.33 (2.49) | 3.43 (2.39)
  Rapid Naming Score | -0.71 (2.46) | 0.21 (2.29)

14. Secondary Outcome: Change From Baseline to Endpoint in CTOPP Composite Score in Participants With ADHD Alone
Description: as for outcome 12
Time Frame: Baseline, 16 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 12 | 9
units on a scale
  Phonological Awareness | 3.66 (2.10) | 7.00 (2.57)
  Phonological Memory | 3.70 (2.61) | 3.48 (2.98)
  Rapid Naming Score | 2.36 (3.01) | 1.63 (3.47)

15. Secondary Outcome: Change From Baseline to Endpoint in Gray Oral Reading Tests-4 (GORT-4) in Participants With Dyslexia Alone
Description: The GORT-4 is a norm-referenced test of oral reading rate, accuracy, fluency, and comprehension valid for individuals aged 6 to 18 years old. The test has two parallel forms, Form A and Form B, that are administered in an alternating fashion (e.g. Week 0-Form A, Week 16-Form B, Week 32-Form A.) with each containing 14 separate stories and 5 multiple-choice comprehension questions for each story. GORT-4 yields the following scores: rate, accuracy, fluency, comprehension, and overall reading ability. Standard scores range from 1-20. Higher scores indicate better reading skills. Lower scores indicate poor reading skills. LS mean was analyzed using LOCF, fixed-effects ANCOVA models of with terms for treatment, gender, baseline, age, treatment*baseline.
Time Frame: Baseline, 16 weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post baseline GORT-4 measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale
  Oral Reading Rate | 0.24 (0.27) | -0.44 (0.27)
  Accuracy | -0.10 (0.46) | -0.72 (0.47)
  Fluency | -0.17 (0.42) | -0.65 (0.42)
  Reading Comprehension | 0.89 (0.77) | -0.29 (0.77)
  Oral Reading Quotient | 2.30 (2.69) | -2.66 (2.72)

16. Secondary Outcome: Change From Baseline to Endpoint in GORT-4 in Participants With ADHD + Dyslexia
Description: The GORT-4 is a norm-referenced test of oral reading rate, accuracy, fluency, and comprehension valid for individuals aged 6 to 18 years old. The test has two parallel forms, Form A and Form B, that are administered in an alternating fashion (e.g. Week 0-Form A, Week 16-Form B, Week 32-Form A.) with each containing 14 separate stories and 5 multiple-choice comprehension questions for each story. GORT-4 yields the following scores: rate, accuracy, fluency, comprehension, and overall reading ability. Standard scores range from 1-20. Higher scores indicate better reading skills. Lower scores indicate poor reading skills. LS mean was analyzed using LOCF, fixed-effects ANCOVA models with terms of treatment, gender, baseline, age, treatment*baseline.
Time Frame: Baseline, 16 weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 12 | 15
units on a scale
  Oral Reading Rate | -0.59 (0.40) | -0.45 (0.37)
  Accuracy | -1.77 (0.53) | -1.02 (0.47)
  Fluency | -1.66 (0.34) | -0.81 (0.31)
  Reading Comprehension | -2.46 (0.67) | -1.55 (0.62)
  Oral Reading Quotient | -14.01 (4.10) | -12.23 (3.40)

17. Secondary Outcome: Change From Baseline to Endpoint in GORT-4 in Participants With ADHD Alone
Description: as for outcome 16
Time Frame: Baseline, 16 weeks
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 12 | 9
units on a scale
  Oral Reading Rate | 0.80 (0.42) | 0.97 (0.48)
  Accuracy | 0.46 (0.35) | -0.17 (0.40)
  Fluency | 0.72 (0.35) | 0.94 (0.40)
  Reading Comprehension | -0.96 (0.59) | 0.79 (0.70)
  Oral Reading Quotient | -0.74 (2.12) | 5.63 (2.46)

18. Secondary Outcome: Change From Baseline to Endpoint Test of Word Reading Efficiency (TOWRE) Total Score in Participants With Dyslexia Alone
Description: The TOWRE is a measure of an individual's ability to pronounce printed words accurately and fluently and is appropriate for individuals aged 6 to 24 years old. The TOWRE contains two subtests: Sight Word Efficiency (SWE) which assesses the number of real printed words that can be accurately identified within 45 seconds and Phonemic Decoding Efficiency (PDE) which measures the number of pronounceable printed non-words that can be accurately decoded within 45 seconds. The total standard score ranges from 35-165. Higher scores indicate higher reading proficiency and lower scores indicate lower reading proficiency. LS mean was calculated using a REML-based, MMRM analysis which includes treatment, baseline, visit, treatment-by-visit interaction, and baseline-by-visit interaction.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post baseline TOWRE measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 14 | 12
units on a scale | 2.21 (1.345) | -0.17 (1.471)

19. Secondary Outcome: Change From Baseline to Endpoint in TOWRE Total Score in Participants With ADHD or ADHD + Dyslexia
Description: as for outcome 18
Time Frame: Baseline, 16 Weeks
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 26 | 28
units on a scale
  ADHD + Dyslexia: number analyzed (Participants) | 13 | 16
  ADHD + Dyslexia | 0.59 (1.435) | 1.18 (1.231)
  ADHD Alone: number analyzed (Participants) | 13 | 12
  ADHD Alone | 4.98 (1.611) | 4.69 (1.844)

20. Secondary Outcome: Change From Baseline to Endpoint in Working Memory Test Battery for Children (WMTB-C) in Participants With Dyslexia Alone
Description: WMTB-C is assessment of working memory capacities, consisting of 9 subtests (Trials Correct Scores [Range from 55-145], Higher scores are better, Lower scores are poor) reflecting 3 main components of working memory: central executive (CE) control/regulation of working memory (Backward Digit Recall, Listening Recall, Counting Recall); phonological loop (PL) responsible for holding verbal information for short periods (Digit Recall, Word List Matching, Word List Recall, Non-word List Recall); and visuo-spatial sketchpad (VSSP) which holds information in visual and spatial form (Block Recall, Mazes Memory). LS mean was analyzed using LOCF, fixed-effects ANCOVA models with terms for treatment, gender, baseline, age, treatment*baseline.
Time Frame: Baseline, 16 Weeks
Population: All randomized participants who received at least one dose of study drug and had evaluable baseline and post baseline WMTB-C measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 14 | 13
units on a scale
  Digit Recall Score | 0.74 (1.25) | 0.94 (1.26)
  Word List Matching Score | 0.34 (2.15) | 0.97 (2.12)
  Word List Recall Score | 0.61 (0.81) | 0.50 (0.83)
  Nonword List Recall Score | -0.10 (0.68) | 0.17 (0.69)
  Block Recall Score | 0.59 (1.23) | 0.82 (1.25)
  Mazes Memory Score | -1.05 (1.87) | -2.96 (1.91)
  Listening Recall Score | 1.41 (0.82) | -0.52 (0.84)
  Counting Recall Score | 1.83 (0.85) | 0.18 (0.88)
  Backward Digit Recall Score | -0.28 (1.52) | 0.65 (1.55)

21. Secondary Outcome: Change From Baseline to Endpoint WMTB-C in Participants With ADHD + Dyslexia
Description: as for outcome 20
Time Frame: Baseline, 16 Weeks
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 12 | 16
units on a scale
  Digit Recall | -0.64 (1.04) | 1.03 (0.93)
  Word List Matching | -0.02 (1.90) | -0.78 (1.72)
  Word List Recall | -0.78 (0.77) | 0.80 (0.70)
  NonWord | 0.12 (0.32) | 1.12 (0.29)
  Block Recall | -1.71 (0.83) | 0.75 (0.77)
  Mazes Memory Score | 3.08 (1.34) | -1.01 (1.22)
  Listening Recall | -0.48 (0.75) | 2.16 (0.68)
  Counting Recall | -2.26 (1.36) | -1.61 (1.21)
  Backward Digit Recall | -0.31 (0.82) | 1.76 (0.74)

22. Secondary Outcome: Change From Baseline to Endpoint WMTB-C in Participants With ADHD Alone
Description: as for outcome 20
Time Frame: Baseline, 16 Weeks
Population: as for outcome 20
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 13 | 10
units on a scale
  Digit Recall | 2.70 (1.76) | 0.94 (1.93)
  Word List Matching | -0.79 (1.61) | 2.03 (1.84)
  Word List Recall | 1.50 (1.06) | 1.17 (1.18)
  NonWord | 1.41 (0.82) | -0.13 (0.90)
  Block Recall | 1.03 (1.36) | 0.44 (1.67)
  Mazes Memory Score | 2.70 (1.61) | 0.16 (1.73)
  Listening Recall | 1.53 (1.06) | 1.57 (1.18)
  Counting Recall | 0.31 (1.02) | -1.02 (1.14)
  Backward Digit Recall | 1.82 (1.23) | 2.15 (1.32)

23. Secondary Outcome: Change From Baseline to Endpoint in BADD-A Total Score in Participants With Dyslexia Alone
Description: The BADD-A is used to assess impairment in executive functions related to ADHD. These include 1) Organizing, prioritizing, and activating to work; 2) Focusing, sustaining and shifting attention to tasks; 3) Regulating alertness, sustaining effort, and processing speed; 4) Managing frustration and modulating emotions; 5) Utilizing working memory and accessing recall (Brown 2001). Scores range from 0-120. The higher the score the more severe the ADD. Scores of 0-39 equate to "ADD possible but not likely". Scores of 40-54 equate to "ADD probable but not certain". Scores of 55-120 equate to "ADD highly probable". LS mean was calculated using a REML-based, MMRM analysis which includes treatment, baseline, visit, treatment-by-visit interaction, and baseline-by-visit interaction.
Time Frame: Baseline, 16 Weeks
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 14 | 13
units on a scale | -7.22 (4.756) | -2.82 (5.022)

24. Secondary Outcome: Change From Baseline to Endpoint in ADHDRS-IV Total Score in Participants With Dyslexia Alone
Description: The ADHDRS-IV-Parent is an 18-item scale with 1 item for each of the 18 symptoms contained in the DSM-IV diagnosis of ADHD. Each item is scored on a 0 to 3 scale: 0=none (never or rarely); 1=mild (sometimes); 2=moderate (often); 3=severe (very often). Total scores range from 0-54. Higher scores indicate higher impairment and lower scores indicate no impairment. LS mean was calculated using a REML-based, MMRM analysis which includes treatment, baseline, visit, treatment-by-visit interaction, and baseline-by-visit interaction.
Time Frame: Baseline, 16 Weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 13 | 12
units on a scale | -1.88 (1.441) | -2.51 (1.492)

25. Secondary Outcome: Change From Baseline to Endpoint in WJ III Individual Scores in Participants With Dyslexia Alone
Description: WJ III (Woodcock et al. 2001) has two parallel forms (A and B) alternating two batteries of tests-Standard and Extended. Standard tests (1 -12) have a broad set of scores. Extended tests (13 -22) have a more in-depth diagnostic assessment of academic strengths and weaknesses. Tests administered were 1, 2, 7, 9, 13, 17, and 20. The standard score scale is a mean (M) of 100 and a standard deviation (SD) of 15. The WJ III ACH has extended standard scores, which is a greater range of standard scores. Scores for each individual test range from 0 to over 200 where 69 and below is very low and 131 and above is very superior. Higher scores indicate better reading skills. LS mean was analyzed using LOCF, fixed-effects ANCOVA models with terms for gender, baseline score, and age.
Time Frame: Baseline, 32 Weeks
Population: All randomized participants who received atomoxetine in both phases and had evaluable baseline and post baseline WJ III measurements. No participants by design were on placebo for both study periods II and III.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 6
units on a scale
  Reading Fluency | 8.96 (3.63)
  Reading Comprehension | 0.24 (1.56)
  Letter Word Identification | 2.12 (1.67)
  Spelling | -1.81 (2.87)
  Spelling of Sounds | 4.67 (4.82)
  Basic Reading Skills | 3.41 (1.72)
  Passage Comprehension Score | 2.17 (5.68)
  Word Attack Score | 5.37 (4.71)
  Reading Vocabulary Score | -2.28 (2.18)

26. Secondary Outcome: Change From Baseline to Endpoint in WJ III Individual Scores in Participants With ADHD + Dyslexia
Description: WJ III (Woodcock et al. 2001) has two parallel forms (A and B) alternating two batteries of tests-Standard and Extended. Standard tests (1 -12) have a broad set of scores. Extended tests (13 -22) have a more in-depth diagnostic assessment of academic strengths and weaknesses. Tests administered were 1, 2, 7, 9, 13, 17, and 20. The standard score scale is a mean (M) of 100 and a standard deviation (SD) of 15. The WJ III ACH has extended standard scores, which is a greater range of standard scores. Scores for each individual test range from 0 to over 200 where 69 and below is very low and 131 and above is very superior. Higher scores indicate better reading skills. LS mean was analyzed using LOCF, fixed-effects ANCOVA models with terms for treatment, gender, baseline score, age, and baseline score by treatment interaction.
Time Frame: Baseline, 32 Weeks
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 5
units on a scale
  Letter Word Identification | 2.40 (3.30)
  Word Attack Score | -0.78 (0.21)
  Reading Vocabulary | 0.71 (1.16)
  Reading Fluency | 2.24 (0.27)
  Reading Comprehension | 2.61 (1.31)
  Spelling | 1.29 (3.68)
  Spelling of Sounds | -1.79 (1.03)
  Basic Reading Skills | 0.70 (0.04)
  Passage Comprehension Score | 3.58 (2.01)

27. Secondary Outcome: Change From Baseline to Endpoint in WJ III Individual Scores in Participants With ADHD Alone
Description: as for outcome 26
Time Frame: Baseline, 32 Weeks
Population: as for outcome 25
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 6
units on a scale
  Letter Word Identification | -1.89 (0.39)
  Word Attack Score | -1.87 (1.73)
  Reading Vocabulary | 5.88 (3.40)
  Reading Fluency | 2.93 (3.82)
  Reading Comprehension | 4.77 (2.39)
  Spelling | 4.04 (2.79)
  Spelling of Sounds | 6.80 (2.79)
  Basic Reading Skills | -2.44 (0.77)
  Passage Comprehension Score | -3.16 (1.09)

28. Secondary Outcome: Change From Baseline to Endpoint in CTOPP Composite Scores in Participants With Dyslexia Alone
Description: as for outcome 12
Time Frame: Baseline, 32 Weeks
Population: All randomized participants who received atomoxetine in both phases and had evaluable baseline and post baseline CTOPP measurements. No participants by design were on placebo for both study periods II and III.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 6
units on a scale
  Phonological Awareness | -0.41 (0.67)
  Phonological Memory | -4.63 (2.41)
  Rapid Naming Score | 3.99 (4.49)

29. Secondary Outcome: Change From Baseline to Endpoint in CTOPP Composite Scores in Participants With ADHD + Dyslexia
Description: as for outcome 12
Time Frame: Baseline, 32 Weeks
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 5
units on a scale
  Phonological Awareness | 12.69 (1.89)
  Phonological Memory | 3.40 (2.27)
  Rapid Naming Score | 4.72 (3.47)

30. Secondary Outcome: Change From Baseline to Endpoint in CTOPP Composite Scores in Participants With ADHD Alone
Description: as for outcome 12
Time Frame: Baseline, 32 Weeks
Population: as for outcome 28
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 6
units on a scale
  Phonological Awareness | 5.90 (6.17)
  Phonological Memory | 5.61 (2.30)
  Rapid Naming Score | 2.67 (0.32)

31. Secondary Outcome: Change From Baseline to Endpoint in GORT-4 in Participants With Dyslexia Alone
Description: The GORT-4 is a norm-referenced test of oral reading rate, accuracy, fluency, and comprehension valid for individuals aged 6 to 18 years old. The test has two parallel forms, Form A and Form B, that are administered in an alternating fashion (e.g. Week 0-Form A, Week 16-Form B, Week 32-Form A.) with each containing 14 separate stories and 5 multiple-choice comprehension questions for each story. GORT-4 yields the following scores: rate, accuracy, fluency, comprehension, and overall reading ability. Standard scores range from 1-20. Higher scores indicate better reading skills. Lower scores indicate poor reading skills. LS mean was analyzed using LOCF, fixed-effects ANCOVA models with terms for treatment, gender, baseline, age, treatment*baseline.
Time Frame: Baseline, 32 Weeks
Population: All randomized participants who received atomoxetine in both phases and had evaluable baseline and post baseline GORT-4 measurements. No participants by design were on placebo for both study periods II and III.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 6
units on a scale
  Oral Reading Rate | 0.63 (0.79)
  Accuracy | -1.93 (0.47)
  Fluency | -0.66 (0.45)
  Reading Comprehension | -0.23 (2.86)
  Oral Reading Quotient | -9.53 (14.45)

32. Secondary Outcome: Change From Baseline to Endpoint in GORT-4 in Participants With ADHD + Dyslexia
Description: as for outcome 31
Time Frame: Baseline, 32 Weeks
Population: as for outcome 31
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 5
units on a scale
  Oral Reading Rate | 0.22 (0.25)
  Accuracy | 0.17 (0.02)
  Fluency | -0.28 (0.34)
  Reading Comprehension | -0.61 (0.31)
  Oral Reading Quotient | -2.23 (1.89)

33. Secondary Outcome: Change From Baseline to Endpoint in GORT-4 in Participants With ADHD Alone
Description: as for outcome 31
Time Frame: Baseline, 32 Weeks
Population: as for outcome 31
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 6
units on a scale
  Oral Reading Rate | 0.05 (0.63)
  Accuracy | -1.44 (0.45)
  Fluency | -0.20 (0.22)
  Reading Comprehension | -0.02 (1.07)
  Oral Reading Quotient | -1.37 (4.86)

34. Secondary Outcome: Change From Baseline to Endpoint in Participants in TOWRE Total Score With Dyslexia Alone
Description: as for outcome 18
Time Frame: Baseline, 32 Weeks
Population: All randomized participants who received atomoxetine in both phases and had evaluable baseline and post baseline TOWRE measurements. No participants by design were on placebo for both study periods II and III.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 15
units on a scale | 3.20 (3.04)

35. Secondary Outcome: Change From Baseline to Endpoint in Participants in TOWRE Total Score With ADHD or ADHD + Dyslexia
Description: as for outcome 18
Time Frame: Baseline, 32 Weeks
Population: as for outcome 34
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 10
units on a scale
  ADHD + Dyslexia: number analyzed (Participants) | 5
  ADHD + Dyslexia | 2.77 (1.99)
  ADHD Alone: number analyzed (Participants) | 5
  ADHD Alone | 6.75 (0.04)

36. Secondary Outcome: Change From Baseline to Endpoint in Participants in WMTB-C With Dyslexia Alone
Description: as for outcome 20
Time Frame: Baseline, 32 Weeks
Population: All randomized participants who received atomoxetine in both phases and had evaluable baseline and post baseline WMTB-C measurements. No participants by design were on placebo for both study periods II and III.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 6
units on a scale
  Digit Recall Score | 0.47 (1.00)
  Word List Matching Score | 1.29 (2.62)
  Word List Recall Score | 0.75 (1.65)
  Nonword List Recall Score | -0.96 (2.45)
  Block Recall Score | 1.25 (2.51)
  Mazes Memory Score | 1.91 (3.74)
  Listening Recall Score | 4.15 (2.14)
  Counting Recall Score | -0.88 (1.39)
  Backwards Digit Recall Score | -0.64 (2.95)

37. Secondary Outcome: Change From Baseline to Endpoint in Participants in WMTB-C With ADHD + Dyslexia
Description: as for outcome 20
Time Frame: Baseline, 32 Weeks
Population: All randomized participants who had received atomoxetine in both phases and had evaluable baseline and post baseline WTMB-C measurements.No participants by design were on placebo for both study periods II and III.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 5
units on a scale
  Digit Recall Score | 0.06 (0.07)
  Word List Matching Score | -4.12 (1.25)
  Word List Recall Score | 3.05 (1.51)
  Nonword List Recall Score | 1.78 (0.42)
  Block Recall Score | 0.56 (1.13)
  Mazes Memory Score | -0.22 (2.73)
  Listening Recall Score | 0.73 (3.37)
  Counting Recall Score | -0.55 (2.47)
  Backward Digit Recall Score | 0.05 (2.95)

38. Secondary Outcome: Change From Baseline to Endpoint in Participants in WMTB-C With ADHD Alone
Description: as for outcome 20
Time Frame: Baseline, 32 Weeks
Population: as for outcome 37
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 5
units on a scale
  Digit Recall Score | 3.75 (0.93)
  Word List Matching Score | -3.37 (0.37)
  Word List Recall Score | 1.25 (0.49)
  Nonword List Recall Score | 1.12 (0.60)
  Block Recall Score | 3.65 (3.48)
  Mazes Memory Score | -1.09 (1.43)
  Listening Recall Score | 4.24 (1.96)
  Counting Recall Score | -3.05 (1.67)
  Backward Digit Recall Score | -0.45 (0.00)

39. Secondary Outcome: Change From Baseline to Endpoint in BADD-A Total Score in Participants With Dyslexia Alone
Description: The BADD-A is used to assess impairment in executive functions related to ADHD. These include 1) Organizing, prioritizing, and activating to work; 2) Focusing, sustaining and shifting attention to tasks; 3) Regulating alertness, sustaining effort, and processing speed; 4) Managing frustration and modulating emotions; 5) Utilizing working memory and accessing recall (Brown 2001). Scores range from 0-120. The higher the score the more severe the ADD. Scores of 0-39 equate to "ADD possible but not likely". Scores of 40-54 equate to "ADD probable but not certain". Scores of 55-120 equate to "ADD highly probable". LS Mean was calculated using ANCOVA model with terms for gender, baseline score, and age.
Time Frame: Baseline, 32 Weeks
Population: All randomized participants who received atomoxetine in both phases and had evaluable baseline and post baseline BADD-A measurements. No participants by design were on placebo for both study periods II and III.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 6
units on a scale | -10.07 (6.70)

40. Secondary Outcome: Change From Baseline to Endpoint in BADD-A Total Score in Participants With ADHD or ADHD + Dyslexia
Description: as for outcome 39
Time Frame: Baseline, 32 Weeks
Population: as for outcome 39
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 11
units on a scale
  ADHD + Dyslexia: number analyzed (Participants) | 5
  ADHD + Dyslexia | -9.44 (7.43)
  ADHD Alone: number analyzed (Participants) | 6
  ADHD Alone | -9.33 (5.04)

41. Secondary Outcome: Change From Baseline to Endpoint in ADHDRS-IV-Parent: Inv Total Score in Participants With Dyslexia Alone
Description: The ADHDRS-IV-Parent is an 18-item scale with 1 item for each of the 18 symptoms contained in the DSM-IV diagnosis of ADHD. Each item is scored on a 0 to 3 scale: 0=none (never or rarely); 1=mild (sometimes); 2=moderate (often); 3=severe (very often). Total scores range from 0-54. Higher scores indicate higher impairment and lower scores indicate no impairment. LS Mean was calculated using ANCOVA model with terms for gender, baseline score, and age.
Time Frame: Baseline, 32 Weeks
Population: All randomized participants who received atomoxetine in both phases and had evaluable baseline and post baseline ADHDRS-IV-Parent: Inv measurements. No participants by design were on placebo for both study periods II and III.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 6
units on a scale | 12.60 (8.17)

42. Secondary Outcome: Change From Baseline to Endpoint in ADHDRS-IV-Parent: Inv Total Score in Participants With ADHD or ADHD +Dyslexia
Description: as for outcome 41
Time Frame: Baseline, 32 Weeks
Population: as for outcome 41
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 11
units on a scale
  ADHD + Dyslexia: number analyzed (Participants) | 5
  ADHD + Dyslexia | -12.96 (2.44)
  ADHD Alone: number analyzed (Participants) | 6
  ADHD Alone | -18.76 (5.89)

43. Secondary Outcome: Change From Baseline to Endpoint in fMRI Activation in Participants With Dyslexia Alone (Pseudoword Rhyming, Semantic-category)
Description: Change From Baseline to Endpoint in fMRI Activation in Participants With Dyslexia Alone (Pseudoword Rhyming, Semantic-category)
Time Frame: From Week 16, Up to Week 32
Population: For this outcome measure, there were no data collected beyond 16 weeks.
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: Change From Baseline to Endpoint in fMRI Activation in Participants With Dyslexia Alone (Stroop Tasks)
Description: Change From Baseline to Endpoint in fMRI Activation in Participants With Dyslexia Alone (Stroop Tasks)
Time Frame: From Week 16, Up to 32 Weeks
Population: Stroop Tasks data were not collected.
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 0 | 0

45. Secondary Outcome: Change From Baseline to Endpoint in fMRI Activation in Participants With ADHD or ADHD + Dyslexia (Pseudoword Rhyming and Semantic-category Tasks)
Description: Change From Baseline to Endpoint in fMRI Activation in Participants With ADHD or ADHD + Dyslexia (Pseudoword Rhyming and Semantic-category Tasks)
Time Frame: From Week 16, Up to Week 32
Population: For this outcome measure, there were no data collected beyond 16 weeks.
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 0 | 0

46. Secondary Outcome: Change From Baseline to Endpoint in fMRI Activation in Participants With ADHD or ADHD + Dyslexia (Stroop Tasks)
Description: Change From Baseline to Endpoint in fMRI Activation in Participants With ADHD or ADHD + Dyslexia (Stroop Tasks)
Time Frame: From Week 16, Up to Week 32
Population: Stroop Tasks data were not collected.
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 0 | 0

47. Secondary Outcome: Change From Baseline to Endpoint in WJ III Individual Scores in Participants With Dyslexia Alone
Description: as for outcome 26
Time Frame: From Week 16, Up to 32 Weeks
Population: All participants who received at least one dose of study drug and had evaluable baseline and post baseline WJ III measurements. The objectives for this portion of the trial centered around participants already exposed to ATX for 16 weeks and therefore no data for PLA/ATX are given.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 6 | 6
units on a scale
  Word Attack Score | 2.79 (2.68) | -1.01 (2.10)
  Letter Word Identification | 2.92 (2.45) | -4.08 (2.02)
  Reading Fluency | 11.03 (3.14) | -1.53 (2.61)
  Reading Comprehension | 4.52 (2.60) | -6.86 (2.16)
  Spelling | -2.90 (3.73) | -1.72 (3.00)
  Spelling of Sounds | 3.33 (3.11) | 0.30 (2.59)
  Basic Reading Skills | 2.87 (1.44) | -3.80 (1.19)
  Passage Comprehension Score | 4.51 (3.30) | -6.92 (2.74)
  Reading Vocabulary Score | 3.02 (2.04) | -4.84 (1.78)

48. Secondary Outcome: Change From Baseline to Endpoint in WJ III Individual Scores in Participants With ADHD + Dyslexia
Description: as for outcome 26
Time Frame: From Week 16, Up to Week 32
Population: as for outcome 47
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 5 | 6
units on a scale
  Word Attack Score | -2.65 (1.81) | -2.62 (1.63)
  Letter Word Identification | 0.50 (3.19) | -1.07 (3.00)
  Reading Vocabulary Score | 0.64 (2.17) | -4.08 (2.08)
  Reading Fluency | 5.46 (2.77) | 6.21 (2.84)
  Reading Comprehension | 0.86 (2.25) | -2.49 (2.07)
  Spelling | 0.45 (2.46) | 0.86 (2.32)
  Spelling of Sounds | -10.17 (3.40) | -3.52 (3.23)
  Basic Reading Skills | -1.29 (1.06) | -2.17 (1.00)
  Passage Comprehension Score | 0.15 (2.06) | 0.52 (1.85)

49. Secondary Outcome: Change From Baseline to Endpoint in WJ III Individual Scores in Participants With ADHD Alone
Description: as for outcome 26
Time Frame: From Week 16, Up to Week 32
Population: as for outcome 47
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 5 | 6
units on a scale
  Word Attack Score | -1.56 (2.06) | -0.58 (1.85)
  Letter Word Identification | -3.89 (4.46) | -1.61 (4.01)
  Reading Vocabulary Score | 5.15 (5.51) | -3.62 (4.26)
  Reading Fluency | 13.05 (2.32) | 4.88 (1.11)
  Reading Comprehension | 3.86 (2.94) | 3.26 (2.67)
  Spelling | 2.07 (4.66) | 1.15 (3.81)
  Spelling of Sounds | -2.65 (3.02) | 2.65 (2.90)
  Basic Reading Skills | -2.70 (3.56) | -1.97 (3.17)
  Passage Comprehension Score | 6.86 (3.42) | 2.31 (3.00)

50. Secondary Outcome: Change From Baseline to Endpoint in CTOPP Composite Scores in Participants With Dyslexia Alone
Description: as for outcome 12
Time Frame: From Week 16, Up to Week 32
Population: All participants who received at least one dose of study drug and had evaluable baseline and post baseline CTOPP measurements. The objectives for this portion of the trial centered around participants already exposed to ATX for 16 weeks and therefore no data for PLA/ATX are given.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 6 | 6
units on a scale
  Phonological Awareness | -1.19 (4.03) | 2.06 (2.82)
  Phonological Memory | -6.96 (3.71) | -1.76 (3.23)
  Rapid Naming Score | 7.24 (5.91) | -2.42 (4.82)

51. Secondary Outcome: Change From Baseline to Endpoint in CTOPP Composite Scores in Participants With ADHD + Dyslexia
Description: as for outcome 12
Time Frame: From Week 16, Up to Week 32
Population: as for outcome 50
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 5 | 6
units on a scale
  Phonological Awareness | 3.54 (1.51) | 5.29 (1.42)
  Phonological Memory | -2.65 (3.34) | 0.12 (2.88)
  Rapid Naming Score | 2.65 (2.02) | 1.21 (1.64)

52. Secondary Outcome: Change From Baseline to Endpoint in CTOPP Composite Scores in Participants With ADHD Alone
Description: as for outcome 12
Time Frame: From Week 16, Up to Week 32
Population: as for outcome 50
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 6 | 5
units on a scale
  Phonological Awareness | -0.33 (2.89) | 9.67 (2.61)
  Phonological Memory | 3.59 (3.37) | 0.84 (3.58)
  Rapid Naming Score | 1.53 (2.36) | 3.51 (2.05)

53. Secondary Outcome: Change From Baseline to Endpoint TOWRE Total Score in Participants With Dyslexia Alone
Description: as for outcome 18
Time Frame: From Week 16, Up to Week 32
Population: All participants who received at least one dose of study drug and had evaluable baseline and post baseline TOWRE measurements. The objectives for this portion of the trial centered around participants already exposed to ATX for 16 weeks and therefore no data for PLA/ATX are given.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 6 | 6
units on a scale | -0.17 (1.808) | 4.17 (1.808)

54. Secondary Outcome: Change From Baseline to Endpoint in TOWRE Total Score in Participants With ADHD or ADHD + Dyslexia
Description: as for outcome 18
Time Frame: From Week 16, Up to Week 32
Population: as for outcome 53
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 10 | 11
units on a scale
  ADHD + Dyslexia: number analyzed (Participants) | 5 | 6
  ADHD + Dyslexia | 3.74 (1.261) | 1.38 (1.151)
  ADHD Alone: number analyzed (Participants) | 5 | 5
  ADHD Alone | 2.03 (4.179) | 1.37 (4.179)

55. Secondary Outcome: Change From Baseline to Endpoint in GORT-4 in Participants With Dyslexia Alone
Description: as for outcome 31
Time Frame: From Week 16, Up to Week 32
Population: All participants who received at least one dose of study drug and had evaluable baseline and post baseline GORT-4 measurements. The objectives for this portion of the trial centered around participants already exposed to ATX for 16 weeks and therefore no data for PLA/ATX are given.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 6 | 6
units on a scale
  Oral Reading Rate | 0.27 (0.43) | -0.64 (0.36)
  Accuracy | 0.40 (0.62) | -0.69 (0.48)
  Fluency | 0.52 (0.67) | -0.64 (0.49)
  Reading Comprehension | 0.06 (1.40) | -0.76 (1.20)
  Oral Reading Quotient | -3.04 (10.51) | -4.91 (8.62)

56. Secondary Outcome: Change From Baseline to Endpoint in GORT-4 in Participants With ADHD+ Dyslexia
Description: as for outcome 31
Time Frame: From Week 16, Up to Week 32
Population: as for outcome 55
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 6 | 6
units on a scale
  Oral Reading Rate | 0.37 (0.73) | 0.31 (0.66)
  Accuracy | 0.07 (0.84) | 0.45 (0.68)
  Fluency | 0.33 (1.15) | 0.52 (1.08)
  Reading Comprehension | 1.75 (1.42) | 3.64 (1.29)
  Oral Reading Quotient | 7.16 (4.57) | 12.92 (4.32)

57. Secondary Outcome: Change From Baseline to Endpoint in GORT-4 in Participants With ADHD Alone
Description: as for outcome 31
Time Frame: From Week 16, Up to Week 32
Population: as for outcome 55
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 6 | 6
units on a scale
  Oral Reading Rate | 0.36 (0.99) | -0.35 (0.70)
  Accuracy | -1.29 (1.00) | 0.15 (0.82)
  Fluency | -0.54 (0.76) | -0.38 (0.57)
  Reading Comprehension | 3.46 (1.05) | -0.04 (0.75)
  Oral Reading Quotient | 8.27 (8.94) | -3.13 (5.38)

58. Secondary Outcome: Change From Baseline to Endpoint in WMTB-C in Participants With Dyslexia Alone
Description: as for outcome 20
Time Frame: From Week 16, Up to Week 32
Population: All randomized participants who received at least one dose of study drug and had baseline and post baseline WMTB-C measurements. The objectives for this portion of the trial centered around participants already exposed to ATX for 16 weeks and therefore no data for PLA/ATX are given.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 6 | 6
units on a scale
  Digit Recall Score | -1.77 (1.78) | 0.45 (1.48)
  Word List Matching Score | 3.98 (4.14) | 1.84 (2.99)
  Word List Recall Score | -0.68 (2.56) | -1.90 (2.27)
  Nonword List Recall Score | 2.25 (0.71) | -0.40 (0.55)
  Block Recall Score | 1.57 (1.55) | -1.73 (1.07)
  Mazes Memory Score | 6.90 (3.29) | 1.27 (2.76)
  Listening Recall Score | 3.44 (1.11) | -1.23 (0.95)
  Counting Recall Score | -2.05 (2.23) | -2.21 (1.87)
  Backward Digit Recall Score | 2.74 (4.47) | 2.49 (2.21)

59. Secondary Outcome: Change From Baseline to Endpoint WMTB-C in Participants With ADHD + Dyslexia
Description: as for outcome 20
Time Frame: From Week 16, Up to Week 32
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 5 | 6
units on a scale
  Digit Recall Score | -1.25 (0.63) | 1.83 (0.59)
  Word List Matching Score | -4.48 (1.74) | -4.40 (1.60)
  Word List Recall Score | 2.34 (0.66) | 2.28 (0.61)
  NonWord List Recall | 2.17 (1.00) | 0.64 (1.57)
  Block Recall Score | -1.71 (2.57) | 3.81 (1.89)
  Mazes Memory Score | -2.82 (2.69) | 1.28 (2.55)
  Listening Recall Score | 1.93 (1.80) | 0.49 (1.45)
  Counting Recall Score | 1.34 (2.52) | -0.89 (2.46)
  Backward Recall Score | 0.76 (2.03) | -0.14 (1.94)

60. Secondary Outcome: Change From Baseline to Endpoint WMTB-C in Participants With ADHD Alone
Description: as for outcome 20
Time Frame: From Week 16, Up to Week 32
Population: as for outcome 58
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 5 | 5
units on a scale
  Digit Recall Score | 2.56 (2.92) | -0.97 (2.19)
  Word List Matching Score | -1.22 (3.84) | -1.71 (3.48)
  Word List Recall Score | -1.23 (1.41) | 1.71 (1.22)
  NonWord List Recall | -1.29 (1.02) | -1.12 (0.87)
  Block Recall Score | -1.14 (1.96) | 0.59 (1.72)
  Mazes Memory Score | 1.11 (2.35) | -2.51 (2.00)
  Listening Recall Score | -1.12 (3.23) | -0.09 (2.94)
  Counting Recall Score | -0.03 (4.53) | -2.90 (3.75)
  Backward Recall Score | -0.68 (2.03) | -0.46 (1.83)

61. Secondary Outcome: Change From Baseline to Endpoint in BADD-A Total Score in Participants With Dyslexia Alone
Description: as for outcome 23
Time Frame: From Week 16, Up to Week 32
Population: All randomized participants who received at least one dose of study drug and had baseline and post baseline BADD-A measurements. The objectives for this portion of the trial centered around participants already exposed to ATX for 16 weeks and therefore no data for PLA/ATX are given.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 6 | 6
units on a scale | -6.96 (5.240) | 7.13 (5.240)

62. Secondary Outcome: Change From Baseline to Endpoint in BADD-A Total Score in Participants With ADHD or ADHD + Dyslexia
Description: as for outcome 23
Time Frame: From Week 16, Up to Week 32
Population: as for outcome 61
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 10 | 11
units on a scale
  ADHD + Dyslexia: number analyzed (Participants) | 5 | 6
  ADHD + Dyslexia | -0.90 (8.646) | 14.59 (7.892)
  ADHD Alone: number analyzed (Participants) | 5 | 5
  ADHD Alone | 1.01 (4.416) | 3.69 (4.461)

63. Secondary Outcome: Change From Baseline to Endpoint in ADHDRS-IV Total Score in Participants With Dyslexia Alone
Description: as for outcome 24
Time Frame: From Week 16, Up to Week 32
Population: All randomized participants who received at least one dose of study drug and had baseline and post baseline ADHDRS-IV measurements. The objectives for this portion of the trial centered around participants already exposed to ATX for 16 weeks and therefore no data for PLA/ATX are given.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 6 | 18
units on a scale | 3.02 (2.537) | 0.27 (1.457)

64. Secondary Outcome: Change From Baseline to Endpoint in ADHDRS-IV-Parent: Inv Total Score in Participants With ADHD or ADHD + Dyslexia
Description: as for outcome 24
Time Frame: From Week 16, Up to Week 32
Population: as for outcome 63
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATX/ATX | ATX/PLA
Number analyzed (Participants) | 10 | 32
units on a scale
  ADHD + Dyslexia: number analyzed (Participants) | 5 | 19
  ADHD + Dyslexia | -0.32 (3.991) | -6.38 (1.946)
  ADHD alone: number analyzed (Participants) | 5 | 13
  ADHD alone | -6.29 (2.546) | -8.83 (1.561)

65. Secondary Outcome: The Number of Participants With Treatment Emergent Adverse Events (TEAE) in Participants With Dyslexia
Description: The number of participants who experienced one or more treatment emergent adverse events (TEAEs) and who had Dyslexia A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: 16 Weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 16 | 15
Participants | 13 | 11

66. Secondary Outcome: The Number of Participants With TEAE in Participants With ADHD or ADHD+Dyslexia.
Description: The number of participants who experienced one or more TEAEs and who had ADHD and ADHD+Dyslexia. A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: 16 Weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 28 | 29
Participants
  ADHD + Dyslexia: number analyzed (Participants) | 15 | 17
  ADHD + Dyslexia | 12 | 14
  ADHD alone: number analyzed (Participants) | 13 | 12
  ADHD alone | 12 | 8

67. Secondary Outcome: The Number of Participants With TEAE in Participants With Dyslexia
Description: The number of participants with at least one TEAE and had Dyslexia. A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: From 16 Weeks Up to Week 32
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ATX/ATX | ATX/PLA | PLA/ATX
Number analyzed (Participants) | 7 | 6 | 12
Participants | 3 | 2 | 8

68. Secondary Outcome: The Number of Participants With TEAE in Participants With ADHD or ADHD+Dyslexia.
Description: The number of participants who experienced one or more TEAEs with ADHD and ADHD + Dyslexia. A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: From Week 16 Up to Week 32
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ATX/ATX | ATX/PLA | PLA/ATX
Number analyzed (Participants) | 12 | 12 | 18
Participants
  ADHD + Dyslexia | 2 | 2 | 10
  ADHD Alone | 3 | 4 | 8

69. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants who had at least one adverse event. A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: 32 Weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Atomoxetine | Placebo | ATX/ATX | ATX/PLA | PLA/ATX
Number analyzed (Participants) | 45 | 44 | 18 | 18 | 35
Participants | 35 | 31 | 8 | 8 | 25

70. Secondary Outcome: Change From Baseline to Endpoint in WJ III Individual Scores in Healthy Participants
Description: WJ III (Woodcock et al. 2001) has two parallel forms (A and B) alternating two batteries of tests-Standard and Extended. Standard tests (1 -12) have a broad set of scores. Extended tests (13 -22) have a more in-depth diagnostic assessment of academic strengths and weaknesses. Tests administered were 1, 2, 7, 9, 13, 17, and 20. The standard score scale is a mean (M) of 100 and a standard deviation (SD) of 15. The WJ III ACH has extended standard scores, which is a greater range of standard scores. Scores for each individual test range from 0 to over 200 where 69 and below is very low and 131 and above is very superior. Higher scores indicate better reading skills.
Time Frame: Baseline, 16 Weeks
Population: All healthy participants who had evaluable baseline and post baseline WJ III measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale
  Letter Word Identification | -3.42 (5.18)
  Word Attack Score | -2.74 (6.54)
  Reading Vocabulary | -0.63 (7.87)
  Reading Fluency | 5.37 (10.45)
  Reading Comprehension | -1.84 (6.98)
  Spelling | 2.21 (5.70)
  Spelling of Sounds | -2.16 (18.35)
  Basic Reading Skills | -3.58 (5.10)
  Passage Comprehension | -2.11 (7.89)

71. Secondary Outcome: Change From Baseline to Endpoint in CTOPP Composite Scores in Healthy Participants
Description: The CTOPP assesses phonological awareness, phonological memory, and rapid naming and is appropriate for ages 7 to 24. The test contains six core subtests. The composite scores are 1) Phonological Awareness, comprised of the standard scores of the Elision and Blending Words; 2) Phonological Memory, comprised of standard scores for Memory for Digits and Non-word Repetition; and 3) Rapid Naming, comprised of standard scores for Rapid Digit Naming and Rapid Letter Naming. Standard scores range from 1-20, and composite scores range from 35-165. Higher scores are better and lower scores are poor.
Time Frame: Baseline, 16 Weeks
Population: All healthy participants who had evaluable baseline and post baseline CTOPP measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale
  Phonological Awareness | 3.63 (11.12)
  Phonological Memory | 2.05 (3.88)
  Rapid Naming Score | 0.63 (10.75)

72. Secondary Outcome: Change From Baseline to Endpoint in GORT-4 in Healthy Participants
Description: The GORT-4 is a norm-referenced test of oral reading rate, accuracy, fluency, and comprehension valid for individuals aged 6 to 18 years old. The test has two parallel forms, Form A and Form B, that are administered in an alternating fashion (e.g. Week 0-Form A, Week 16-Form B, Week 32-Form A.) with each containing 14 separate stories and 5 multiple-choice comprehension questions for each story. GORT-4 yields the following scores: rate, accuracy, fluency, comprehension, and overall reading ability. Standard scores range from 1-20. Higher scores indicate better reading skills. Lower scores indicate poor reading skills.
Time Frame: Baseline, 16 weeks
Population: All healthy participants who had evaluable baseline and post baseline GORT-4 measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale
  Oral Reading Rate | 0.74 (1.52)
  Accuracy | 0.68 (2.60)
  Fluency | 0.74 (1.97)
  Reading Comprehension | -0.16 (2.95)
  Oral Reading Quotient | -3.42 (24.58)

73. Secondary Outcome: Change From Baseline to Endpoint TOWRE Total Score in Healthy Participants
Description: The TOWRE is a measure of an individual's ability to pronounce printed words accurately and fluently and is appropriate for individuals aged 6 to 24 years old. The TOWRE contains two subtests: Sight Word Efficiency (SWE) which assesses the number of real printed words that can be accurately identified within 45 seconds and Phonemic Decoding Efficiency (PDE) which measures the number of pronounceable printed non-words that can be accurately decoded within 45 seconds. The total standard score ranges from 35-165. Higher scores indicate higher reading proficiency and lower scores indicate lower reading proficiency. LS mean was calculated using a REML-based, MMRM analyses which includes diagnostic group, visit, and diagnostic group-by-visit interaction.
Time Frame: Baseline, 16 Weeks
Population: All healthy participants who had evaluable baseline and post baseline TOWRE measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale | 0.20 (1.487)

74. Secondary Outcome: Change From Baseline to Endpoint in WMTB-C in Healthy Participants
Description: WMTB-C is assessment of working memory capacities, consisting of 9 subtests (Trials Correct Scores [Range from 55-145], Higher scores are better, Lower scores are poor) reflecting 3 main components of working memory: central executive (CE) control/regulation of working memory (Backward Digit Recall, Listening Recall, Counting Recall); phonological loop (PL) responsible for holding verbal information for short periods (Digit Recall, Word List Matching, Word List Recall, Non-word List Recall); and visuo-spatial sketchpad (VSSP) which holds information in visual and spatial form (Block Recall, Mazes Memory).
Time Frame: Baseline, 16 Weeks
Population: All healthy participants who had evaluable baseline and post baseline WMTB-C measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale
  Digit Recall Score | 2.47 (4.50)
  Word List Matching Score | -0.95 (5.38)
  Word List Recall Score | 1.79 (2.53)
  Nonword List Recall Score | 0.58 (4.31)
  Block Recall Score | 1.63 (4.83)
  Mazes Memory Score | 1.11 (7.72)
  Listening Recall Score | -0.58 (3.61)
  Counting Recall Score | 0.37 (3.44)
  Backward Digit Recall Score | 2.95 (4.17)

75. Secondary Outcome: Change From Baseline to Endpoint in BADD-A Total Score in Healthy Participants
Description: The BADD-A is used to assess impairment in executive functions related to ADHD. These include 1) Organizing, prioritizing, and activating to work; 2) Focusing, sustaining and shifting attention to tasks; 3) Regulating alertness, sustaining effort, and processing speed; 4) Managing frustration and modulating emotions; 5) Utilizing working memory and accessing recall (Brown 2001). Scores range from 0-120. The higher the score the more severe the ADD. Scores of 0-39 equate to "ADD possible but not likely". Scores of 40-54 equate to "ADD probable but not certain". Scores of 55-120 equate to "ADD highly probable". LS mean was calculated using a REML-based, MMRM analysis which includes the effects of diagnostic group, visit, and diagnostic group-by-visit interaction.
Time Frame: Baseline, 16 Weeks
Population: All participants who had evaluable baseline and post baseline BADD-A measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale | 1.42 (3.572)

76. Secondary Outcome: Change From Baseline to Endpoint in ADHDRS-IV Total Score in Healthy Participants
Description: The ADHDRS-IV-Parent is an 18-item scale with 1 item for each of the 18 symptoms contained in the DSM-IV diagnosis of ADHD. Each item is scored on a 0 to 3 scale: 0=none (never or rarely); 1=mild (sometimes); 2=moderate (often); 3=severe (very often). Total scores range from 0-54. Higher scores indicate higher impairment and lower scores indicate no impairment. LS mean was calculated using a REML-based, MMRM analysis which includes diagnostic group, visit, and diagnostic group-by-visit interaction.
Time Frame: Baseline, 16 Weeks
Population: All healthy participants who had evaluable baseline and post baseline ADHDRS-IV measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale | 0.15 (1.055)

77. Secondary Outcome: Change From Baseline to Endpoint in WJ III Individual Scores in Healthy Participants
Description: as for outcome 70
Time Frame: Baseline, 32 Weeks
Population: All healthy participants who had baseline and post-baseline WJ III measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale
  Letter Word Identification | -0.37 (5.45)
  Word Attack Score | -3.58 (7.23)
  Reading Vocabulary | 0.79 (7.79)
  Reading Comprehension | 0.47 (7.99)
  Reading Fluency | 7.84 (11.69)
  Spelling | 1.95 (4.49)
  Spelling of Sounds | 3.63 (18.94)
  Basic Reading Skills Score | -2.00 (5.35)
  Passage Comprehension | 0.05 (9.34)

78. Secondary Outcome: Change From Baseline to Endpoint in CTOPP Composite Scores in Healthy Participants
Description: as for outcome 71
Time Frame: Baseline, 32 weeks
Population: All healthy participants who had evaluable baseline and post baseline CTOPP measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale
  Phonological Awareness | 3.63 (11.12)
  Phonological Memory | 2.05 (3.88)
  Rapid Naming Score | 0.63 (10.75)

79. Secondary Outcome: Change From Baseline to Endpoint in GORT-4 in Healthy Participants
Description: as for outcome 72
Time Frame: Baseline, 32 Weeks
Population: All healthy participants who had evaluable baseline and post baseline GORT-4 measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale
  Oral Reading Rate | 0.74 (1.52)
  Accuracy | 0.68 (2.60)
  Fluency | 0.74 (1.97)
  Comprehension | -0.16 (2.95)
  Oral Reading Quotient | -3.42 (24.58)

80. Secondary Outcome: Change From Baseline to Endpoint in TOWRE Total Score in Healthy Participants
Description: The TOWRE is a measure of an individual's ability to pronounce printed words accurately and fluently and is appropriate for individuals aged 6 to 24 years old. The TOWRE contains two subtests: Sight Word Efficiency (SWE) which assesses the number of real printed words that can be accurately identified within 45 seconds and Phonemic Decoding Efficiency (PDE) which measures the number of pronounceable printed non-words that can be accurately decoded within 45 seconds. The total standard score ranges from 35-165. Higher scores indicate higher reading proficiency and lower scores indicate lower reading proficiency. LS mean was calculated using a REML-based, MMRM analysis which includes diagnostic group, visit, and diagnostic group-by-visit interaction.
Time Frame: Baseline, 32 Weeks
Population: All healthy participants who had evaluable baseline and post baseline TOWRE measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale | 4.05 (1.578)

81. Secondary Outcome: Change From Baseline to Endpoint in WMTB-C in Healthy Participants
Description: as for outcome 74
Time Frame: Baseline, 32 Weeks
Population: All healthy participants who had evaluable baseline and post baseline WMTB-C measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale
  Digit Recall Score | 2.47 (4.50)
  Word List Matching Score | -0.95 (5.38)
  Word List Recall Score | 1.79 (2.53)
  Nonword List Recall Score | 0.58 (4.31)
  Block Recall Score | 1.63 (4.83)
  Mazes Memory Score | 1.11 (7.72)
  Listening Recall Score | -0.58 (3.61)
  Counting Recall Score | 0.37 (3.44)
  Backwards Digit Recall Score | 2.95 (4.17)

82. Secondary Outcome: Change From Baseline to Endpoint in BADD-A Total Score in Healthy Participants
Description: The BADD-A is used to assess impairment in executive functions related to ADHD. These include 1) Organizing, prioritizing, and activating to work; 2) Focusing, sustaining and shifting attention to tasks; 3) Regulating alertness, sustaining effort, and processing speed; 4) Managing frustration and modulating emotions; 5) Utilizing working memory and accessing recall (Brown 2001). Scores range from 0-120. The higher the score the more severe the ADD. Scores of 0-39 equate to "ADD possible but not likely". Scores of 40-54 equate to "ADD probable but not certain". Scores of 55-120 equate to "ADD highly probable". LS mean was calculated using a REML-based, MMRM which includes the effects of diagnostic group, visit, diagnostic group-by-visit interaction.
Time Frame: Baseline, 32 Weeks
Population: All healthy participants who had evaluable baseline and post baseline BADD-A measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale | 5.74 (3.991)

83. Secondary Outcome: Change From Baseline to Endpoint in ADHDRS-IV-Parent: Inv Total Score in Healthy Participants
Description: The ADHDRS-IV-Parent is an 18-item scale with 1 item for each of the 18 symptoms contained in the DSM-IV diagnosis of ADHD. Each item is scored on a 0 to 3 scale: 0=none (never or rarely); 1=mild (sometimes); 2=moderate (often); 3=severe (very often). Total scores range from 0-54. Higher scores indicate higher impairment and lower scores indicate no impairment. LS mean was calculated using a REML-based, MMRM analysis which includes the effects of diagnostic group, visit, diagnostic group-by-visit interaction.
Time Frame: Baseline, 32 Weeks
Population: All healthy participants who had evaluable baseline and post baseline ADHDRS-IV measurements.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Healthy Participants
Number analyzed (Participants) | 19
units on a scale | 1.17 (1.046)

ADVERSE EVENTS:
Time Frame: Baseline Up To 34 Weeks
Description: The safety population includes all randomized participants who received one dose of study drug. Healthy participants did not receive any drug.
Groups:
- Atomoxetine: Atomoxetine 1.0 to 1.4 mg/kg was administered orally once daily in the morning for 16 weeks, during SP II. All eligible participants who received atomoxetine during SP II and completed that period were re-randomized to atomoxetine or placebo in SP III.
Arm/Group | Atomoxetine | Placebo | ATX/ATX | ATX/PLA | PLA/ATX
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44 | 0/18 | 0/18 | 0/35
Other Adverse Events (participants affected / at risk) | 35/45 | 31/44 | 8/18 | 8/18 | 25/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Atomoxetine (N=45) | Placebo (N=44) | ATX/ATX (N=18) | ATX/PLA (N=18) | PLA/ATX (N=35)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 10 (10) | 12 (12) | 0 (0) | 0 (0) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 15 (15) | 5 (5) | 0 (0) | 1 (1) | 3 (3)
Therapeutic response unexpected (General disorders) | 13 (20) | 10 (12) | 2 (2) | 3 (5) | 5 (6)
Influenza (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 9 (9)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 2 (2) | 0 (0) | 0 (0) | 8 (8)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 12 (12) | 6 (6) | 0 (0) | 0 (0) | 3 (3)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Emotional disorder (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Irritability (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/18 (0) | 0/17 (0) | 0/4 (0) | 0/10 (0) | 1/12 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Educational problem (Social circumstances) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less